CLINICAL TRIAL: NCT05776706
Title: Clinical Trial for the Evaluation of the Accuracy of Augmented Reality Based Neuronavigation System
Brief Title: Clinical Trial for the Validation of AR Based Neuronavigation System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chul-Kee Park, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SNUH-AR001
Record Dates: First submitted 2022-12-05; First posted 2023-03-20 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Brain Neoplasms; Cerebral Aneurysm; Cerebral Arteriovenous Malformation; Navigation, Spatial
Keywords: augmented reality; neuronavigation; brain neoplasms; cerebral arteriovenous malformation; cerebral aneurysm
MeSH Terms: conditions — Brain Neoplasms; Intracranial Aneurysm; Intracranial Arteriovenous Malformations; Spatial Navigation

STUDY DESIGN:
Intervention Model Description: Patients who undergo craniotomy using navigation system for cerebral disease in a single institution
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): We will set up 2 navigation systems, newly developed AR-based navigation and conventional navigation system, to surgeries of all participants.
  Surgeons will perform all surgical planning and operations with reference to the conventional navigation system. In this process, the errors of the existing navigation and the newly developed navigation will be measured and compared in 3D at several points, and the points are as follows:
  1. Fiducial markers
  2. Nasion
  3. Tumor's margin (anterior, posterior, superior, inferior)
  Interventions: Diagnostic Test: AR-based navigation

INTERVENTIONS:
Diagnostic Test: AR-based navigation — The surgeon will perform all surgical planning and operations with reference to the existing navigation. In this process, the errors of the existing navigation and the newly developed navigation are measured and compared in 3D at several points, and the points are as follows.
  1. Fiducial markers
  2. Nasion
  3. Tumor's margin (anterior, posterior, superior, inferior)

SUMMARY:
The goal of this clinical trial is to test augmented reality (AR) based neuronavigation system in surgeries for patients of brain neoplasm or cerebral vascular disease. The main questions it aims to answer are:

• AR based neuronavigation system can achieve accuracy that is not inferior to conventional intraoperative navigation system.

Participants will participate the study after informed consent. When participants undergo surgery for their brain tumor, we will set up 2 types of neuronavigation, conventional navigation system and developed AR based neuronavigation system. Surgeon will plan and conduct surgery based on only conventional navigation system, but 3D errors at several selected points between two types of navigation will be measured and analyzed.

DETAILED DESCRIPTION:
Being developed AR navigation were reported in our following papers:

1. Dho YS, et al., Development of an inside-out augmented reality technique for neurosurgical navigation. Neurosurgical Focus. 2021 Aug 1;51(2):E21. (doi.org/10.3171/2021.5.FOCUS21184)
2. Moon HC, et al., Navigation of frameless fixation for gamma knife radiosurgery using fixed augmented reality. Scientific Reports. 2022 Mar 16;12(1):1-0. (doi.org/10.3171/2021.5.FOCUS21184)

This study aims to evaluate the accuracy of anatomical localization of a newly developed augmented reality-based neurosurgery navigation. After 3-dimensional (3D) modeling of the brain of a patient with brain tumor or cerebral vascular disease through 3D image segmentation extraction and modeling, the Augmented Reality (AR)-based navigation developed by this research team can be used with a commercially available visualization device, such as iPad, iPhone, and Hololens2, to evaluate the accuracy.

The AR-based navigation obtained approval from the Ministry of Food and Drug Safety of Republic of Korea (class 2 medical device) in February 2022. Through this clinical tria that compare accuracy with existing conventional intraoperative neuronavigation system, we will evaluate whether it shows equivalent performance to replace the existing navigation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older who underwent MRI or CT scan due to brain tumor or cerebrovascular disease
* Adult patients aged 18 years or older who need surgical treatment using navigation for brain tumor or cerebrovascular disease

Exclusion Criteria:

* Cases where application of navigation is not necessary according to the judgment of the researcher or surgeon
* When the patient or guardian does not agree
* Patients with anatomical deformation due to previous surgery or requiring emergency surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The degree of 3-dimensional error at each measurement points (mm) | 6 hours
  Fiducial markers, nasion
The degree of 3-dimensional error at each measurement points (mm) after durotomy | 6 hours
  Tumor's margin, ICA bifurcation, et al.

SECONDARY OUTCOMES:
Non-inferiority of AR-based navigation compared to conventional navigation | 12 months
  Statistical comparison of the average value between the error with the actual position of conventional navigation and the error with the actual position of AR navigation.
Time required to set up and use each navigation | 6 hours
  Time required to match conventional navigation and AR navigation, respectively.
Economic analysis for each navigation | 12 months
  Economic benefits that can be expected if AR-based navigation can replace conventional navigation will be assessed. Cost for surgery, cost of whole admission period, and hospital day will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Kee Park, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No